CLINICAL TRIAL: NCT03423810
Title: Assessing a Dose-Response Relationship of Hydralazine and Its Effects on DNA Methyltransferase 1 in Polycystic Kidney Disease Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00141337; UL1TR002366 (NIH)
Record Dates: First submitted 2018-01-31; First posted 2018-02-06 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Polycystic Kidney Diseases
MeSH Terms: conditions — Polycystic Kidney Diseases | interventions — Hydralazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Group 1: Hydralazine (Experimental): Participants will take hydralazine twice daily for total of 6 weeks. The dose of hydralazine will be increased every 2 weeks.
  Interventions: Drug: Hydralazine

INTERVENTIONS:
Drug: Hydralazine — Participants will be asked to take pills two times per day for 6 weeks. This is a dose increasing study with potential doses ranging from 5 mg two times per day to 50 mg two times per day.

SUMMARY:
The purpose of this study is to find a protein (ex. Polycystin 1 or mucin and cadherin like protein) in the urine that is changed after treatment of hydralazine.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of ADPKD
* estimated glomerular filtration rate (eGFR) > 60 ml/min/1.73m^2

Exclusion Criteria:

* History of systemic lupus erythematous or other rheumatologic disorder
* Baseline anti-nuclear antibody (ANA) >1:80 for females and >1:40 for males
* Blood pressure < 120/80 without anti-hypertensive
* Angina pectoris or myocardial infarction in the last 6 months
* Liver disease
* Allergy to hydralazine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Change in polycystin-1 (PC1) | Change from Baseline to Week 8
Change in mucin-like protocadherin (MUPCDH) | Change from Baseline to Week 8

SECONDARY OUTCOMES:
Circulating methylated RASAL1 levels | Change from Baseline to Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Kerri McGreal, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States